CLINICAL TRIAL: NCT00138632
Title: A Randomized, Double-Masked, Multicenter, Phase I/II Study of the Safety of PTK787 Administered to Patients With Predominantly Classic , Minimally Classic or Occult With no Classic Subfoveal Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: Safety and Efficacy of Oral PTK787 in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-Related Macular Degeneration (AMD)
Acronym: ADVANCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPTK787E2201
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Wet Age-Related Macular Degeneration
Keywords: Wet Age-related macular degeneration; PTK787
MeSH Terms: interventions — vatalanib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: PTK787
- 2 (Experimental)
  Interventions: Drug: PTK787
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTK787 — Visudyne® + PTK787, 500 mg/day
  Arms: 1
Drug: PTK787 — Visudyne® + PTK787 1000 mg/day
  Arms: 2
Drug: Placebo — Visudyne® + Placebo
  Arms: 3

SUMMARY:
This study evaluates the tolerability and safety of 3 months treatment with PTK787 tablets given daily. It also explores the efficacy of the compound in patients with wet age-related macular edema.

In Cohort 1 verteporfin/PDT is the active control. The protocol was amended to reflect the current standard of care for AMD. As a result, ranibizumab is the active control for Cohort 2.

ELIGIBILITY:
Inclusion criteria

* Male ≥ 65 years old or female ≥ 50 years old, with aged related macular degeneration
* Patients with subfoveal choroidal neovascularization secondary to AMD

Exclusion criteria

* Eye disease that may result in visual loss during the study
* Uncontrolled high blood pressure, despite chronic stable treatment: systolic ≥ 140 mmHg, Diastolic ≥ 90 mmHg
* Chronic therapy with topical, local or systemic corticosteroids.
* Use of other investigational drugs within 30 days
* Pregnant or nursing (lactating) women.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by visual acuity measurements, ophthalmic examinations, vital signs, laboratory assessments, and adverse events up to 12 months | up to 12 months

SECONDARY OUTCOMES:
Change in macular edema from Baseline up to Month 3 Change in best-corrected visual acuity (BCVA) from Baseline up to Month 3 Change in size of fluorescein leakage Baseline up to Month 3 | from baseline up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — Novartis
Locations (11):
- United States (7):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Porter Adventist Hospital, Eye Lab, Denver, Colorado
  - USF Eye Institute, Tampa, Florida
  - Springfield Clinic, LLP, Springfield, Illinois
  - Wilmer Eye Institute, Baltimore, Maryland
  - Lahey Clinic Medical Center, Eye institute, Peabody, Massachusetts
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
- Australia (4):
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigational Site, Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, East Melbourne, Victoria